CLINICAL TRIAL: NCT01720550
Title: PG2 Treatment for Improving Fatigue Among Advanced Cancer Patients Under Standard Palliative Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PH-CP012 (II)
Record Dates: First submitted 2012-10-29; First posted 2012-11-02 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Cancer-related Fatigue
Keywords: Cancer-related fatigue; Palliative Treatment; Astragalus polysaccharides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PG2 High Dose (Experimental): Astragalus Polysaccharides 500 mg
  Interventions: Drug: Astragalus Polysaccharides 500 mg
- PG2 Low Dose (Experimental): Astragalus Polysaccharides 250 mg
  Interventions: Drug: Astragalus Polysaccharides 250 mg

INTERVENTIONS:
Drug: Astragalus Polysaccharides 500 mg — PG2 (500 mg in 500 ml saline), t.i.w. via i.v. infusion for 2.5-3.5 hours over 2 treatment cycles (8 weeks)
  Other Names: PG2 Injection 500 mg
  Arms: PG2 High Dose
Drug: Astragalus Polysaccharides 250 mg — PG2 (500 mg in 500 ml saline), t.i.w. via i.v. infusion for 2.5-3.5 hours over 2 treatment cycles (8 weeks)
  Other Names: PG2 Injection 250 mg
  Arms: PG2 Low Dose

SUMMARY:
The objective of this study is to conduct a trial in the spirit of providing as much as possible the benefit of PG2 treatment to eligible patients and to evaluate the efficacy and safety of different doses of PG2 treatment for relieving fatigue among advanced cancer patients who are under standard palliative care (SPC) at hospice setting and have no further curative options available. Patient's fatigue status, to be measured by the Brief Fatigue Inventory-Taiwanese Form (BFI-T), will be the primary endpoint. The fatigue improvement response rate among patients between two study arms will then be compared as the basis for efficacy evaluation at the end of the first treatment cycle, and will be the primary endpoint. Other endpoints, the fatigue improvement response rate and the mean fatigue scores change from baseline among patients within and between cycles will be included in the secondary efficacy endpoints, and will be compared between two study arms. Patients' quality of sleep, appetite, pain, fatigue, nausea, vomiting and global quality of life (QoL) will be also measured by 11 questions (SS11) from EORTC(European Organization) for Research and Treatment of Cancer QLQ-C30 for secondary endpoint evaluation. The other secondary endpoints include Karnofsky performance scores, and weight change and its related c-reactive protein level of the patients.

DETAILED DESCRIPTION:
This is a trial to evaluate use of different doses of PG2 treatment for fatigue improvement in advanced cancer patients who are under standard palliative care at hospice setting and have no further curative options available. Only patients who give consent to participate in this study and meet all other inclusion and exclusion criteria will be eligible to enroll into this study. All patients will continue the standard palliative care (SPC) during this study.

The main aim of this trial is to compare improvement of patient's fatigue status between patients with different doses of PG2 treatment. Patient's fatigue status will be assessed by the Brief Fatigue Inventory-Taiwanese (BFI-T) Form. Each patient's fatigue improvement response will be defined as an improvement in the mean fatigue scores by at least 10% from baseline. Other quality of life parameters will be measured by the 11 questions (SS11) of the EORTC QLQ-C30 and by Karnofsky performance scale. Patient's weight change and its related c-reactive protein will be followed. There are two study arms in this trial: 1) the PG2 High Dose arm; and 2) the PG2 Low Dose arm.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form
* ≧ 20 years old
* Have locally advanced or metastatic cancer or inoperable advanced cancer
* Under standard palliative care (SPC) at hospice setting and have no further curative options available
* BFI score ≧ 4
* Life expectancy of at least 3 months as determined by the investigator
* Willing and able to complete quality of life questionnaires

Exclusion Criteria:

* Pregnant or breast-feeding
* Uncontrolled systemic disease
* Take central nervous system stimulators within 30 days before screening
* Have enrolled or have not yet completed other investigational drug trials within 30 days before screening
* Karnofsky Performance Scores less than 30 %
* Diagnosed as dying status

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Fatigue Improvement Response Rate | 4 weeks
  Patient's fatigue status will be measured by the Brief Fatigue Inventory-Taiwanese Form (BFI-T). The fatigue improvement response rate among patients between two study arms will be compared as the basis for efficacy evaluation at the end of the first treatment cycle (4th week).

SECONDARY OUTCOMES:
The fatigue improvement response rate among patients within and between cycles (by BFI-T) | 8 weeks
The fatigue improvement by multiple BFI-T score percentage change levels among patients between two study arms | 8 weeks
The mean of patients' fatigue score change from baseline within and between cycles (by BFI-T) | 8 weeks
Symptoms and Quality of Life Assessments: SS11 from EORTC QLQ-C30 (including the evaluation of the quality of sleep, appetite, pain, fatigue, nausea, vomiting and global quality of life) | 8 weeks
Karnofsky performance score | 8 weeks
The correlation between Weight change and the related blood c-reactive protein level | 8 weeks
Physical Examination | 8 weeks
Labolatory Safety Examination | 8 weeks
  Included hematological, biochemical and urine examination
Incidence of Adverse Events as a Measure of Safety and Tolerability | 8 weeks
Vital signs | 8 weeks
Immune Biomarkers | 8 weeks
  This outcome specified for academic research was designed in add-on protocol (only submitted to IRB)

CONTACTS AND LOCATIONS:
Overall Officials: Yuen-Liang YL Lai, MD, Principal Investigator — Mackay Memorial Hospital
Locations (9):
- Taiwan (9):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital, Kaohsiung Branch, Kaohsiung City
  - Chang Gung Memorial Hospital, Lovers Lake Branch, Keelung
  - China Medical University Hospital, Taichung
  - Chi Mei Hospital, Loiuying Campus, Tainan
  - Mackay Memorial Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Medical University -Shung Ho Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided